CLINICAL TRIAL: NCT07341308
Title: Does Vitamin C Increase the Body Heat Generated By The Nervous System?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 6115
Record Dates: First submitted 2025-12-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metabolism Changes; Vitamin D
Keywords: isoproterenol; vitamin c; vitamin d; body temperature
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Response to beta-adrenergic stimulation without vitamin C (No Intervention): Isoproterenol will be infused with saline only
- Adding vitamin C to beta-adrenergic receptor stilmulation (Experimental): Isoproterenol will be infused with vitamin C
  Interventions: Other: Vitamin C

INTERVENTIONS:
Other: Vitamin C — Vitamin C will be co-infused with isoproterenol
  Arms: Adding vitamin C to beta-adrenergic receptor stilmulation

SUMMARY:
The goals of this clinical trial are to determine whether or not vitamin C is able to: (1) increase the body heat generated by the sympathetic nervous system; and, (2) increase circulating vitamin D concentration during sympathetic nervous system stimulation in adult humans aged 18-40 years who meet the criteria for overweight based on body mass index. The main question it aims to answer are:

1. By how much does body temperature increase during stimulation of beta-adrenergic receptors when vitamin C is given.
2. By how much does circulating vitamin D concentration increase during stimulation of beta-adrenergic receptors when vitamin C is given.

Participants will will be asked to:

* undergo measures of body temperature
* have blood sampled on two separate occasions: once during stimulation of beta adrenergic receptors, and once during stimulation of beta-adrenergic receptors while also been given vitamin C.

DETAILED DESCRIPTION:
Participants will be required to visit the lab twice. During each visit, beta-adrenergic receptors will be stimulated with isoproterenol. The two visits are identical in every way with one exception: during one visit the isoproterenol will be delivered with saline only, and during the other visit the isoproterenol will be delivered with saline and vitamin C. The order of the visits will be randomized. Body temperature will be measured with a thermometer and a thermal camera. venous blood will be sampled and circulating vitamin D concentration will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years (inclusive)
* Body mass index greater than or equal to 25 kg/m2 and less than 30 kg/m2
* Weight stable (no change in body mass greater than 5 Lbs. within the previous 6 months.
* Willing to abstain from caffeine and alcohol for 24-hours prior to two different study visits
* Competency in English as assessed by comprehension of the Informed Consent. This is study involves invasive procedures and infusion of a systemic vasoactive agent (isoproterenol); for safety reasons, the ability for clear and rapid communication will be necessary between the research participants and the investigators.

Exclusion Criteria:

* History of autonomic, cardio-pulmonary, and/or metabolic disease (including heart failure, hypertension, arrhythmia, vascular disease, and/or diabetes)
* Pregnancy or breast feeding
* Habitual use of tobacco/nicotine products or recreational drugs (2 or more uses within the previous month)
* History of a "sulfite allergy" as it is a relative contraindication to isoproteronol use.
* Has ingested vitamin supplements and/or antioxidant supplements during the previous 4-weeks (e.g. Vitamin C, Vitamin E, Multi-vitamins, etc.)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-12-08 (Estimated)

PRIMARY OUTCOMES:
Body Temperature | Prior to and immediately after a dose of isoproterenol. This corresponds to 0 minutes (baseline) and immediately after each dose of isoproterenol at minutes 30, 60 and 90.
  Body temperature will be measured using an oral thermometer
Vitamin D | Prior to and immediately after a dose of isoproterenol. This corresponds to 0 minutes (baseline) and immediately after each dose of isoproterenol at minutes 30, 60 and 90.
  Circulating vitamin D concentration

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bell, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No